CLINICAL TRIAL: NCT06997380
Title: Assessment of the Safety and Efficacy of the DensiStim Medical Device, an Injectable Liposomal Gel, in Adult Participants
Brief Title: Evaluation of the Safety and Efficacy of an Injectable Liposomal Gel
Acronym: DensiStim
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Biovico Sp. z o.o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DensiStim
Record Dates: First submitted 2025-05-14; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Skin Aging; Skin Wrinkling; Facial Skin Laxity; Facial Wrinkles
Keywords: hyaluronic acid; skin biostimulation; intradermal injection; facial skin rejuvenation; dry skin; thin skin; skin rejuvenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- needle group (Experimental): product administration using a needle
  Interventions: Device: Injection of the investigational product via needle; Procedure: Clinical assessment; Procedure: Ultrasound measurement; Procedure: Multispectral imaging
- cannula group (Experimental): product administration using a cannula
  Interventions: Device: Injection of the investigational product via cannula; Procedure: Clinical assessment; Procedure: Ultrasound measurement; Procedure: Multispectral imaging

INTERVENTIONS:
Device: Injection of the investigational product via needle — A hyaluronic acid solution (concentration 2.2%) with the addition of lecithin in the form of liposomes (concentration 0.08%) via needle
  Arms: needle group
Device: Injection of the investigational product via cannula — A hyaluronic acid solution (concentration 2.2%) with the addition of lecithin in the form of liposomes (concentration 0.08%) via cannula
  Arms: cannula group
Procedure: Clinical assessment — Clinical assessment of facial skin condition
Procedure: Ultrasound measurement — Ultrasound measurement of facial skin thickness
Procedure: Multispectral imaging — Multispectral imaging and analysis of facial skin

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of intradermal injections of the medical device - hyaluronic acid with the addition of lecithin - in a population of participants with thin, dry, and sagging facial skin.

DETAILED DESCRIPTION:
A total of 36 participants are planned to be enrolled in the study (18 in each group: Group 1 - product administration using a needle; Group 2 - product administration using a cannula).

The primary endpoint will be the change in facial skin thickness resulting from three administrations of the DensiStim product, assessed no later than 8 weeks after the last procedure, based on ultrasound (US) measurements. Ultrasound measurements will also be compared between visits and between study arms.

Changes in aesthetic improvement will be assessed by both the participant and the Investigator. The safety of the investigational medical device will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Female sex;
2. Age over 18 years;
3. Caucasian race;
4. Thin, dry, and sagging facial skin;
5. Signing an informed consent form;
6. Commitment to refrain from undergoing facial therapies that may affect skin condition;
7. Negative pregnancy test result and commitment to use a contraceptve method;

Exclusion Criteria:

1. Scars, birthmarks, or tattoos on the face that could interfere with the assessment of skin condition;
2. Presence of open wounds, ulcers, active infections, or other significant skin damage at the planned injection site;
3. Receipt of intradermal facial injections with native hyaluronic acid, platelet-rich plasma, or other injectable therapies within 6 months prior to study initiation;
4. Receipt of intradermal facial injections with slowly absorbable or non-absorbable filler products within 12 months prior to study initiation;
5. Known hypersensitivity to any component of the investigational product;
6. Dermatitis or dermatological disease of inflammatory and/or infectious nature at the planned injection site;
7. History of cancer, autoimmune disease, or immunodeficiency;
8. Use of medications affecting blood coagulation;
9. Use of topical antihistamines, corticosteroids, or retinoids on the face within 4 weeks prior to the study;
10. Pregnancy or breastfeeding;
11. Participation or planned participation in other clinical trials;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-05-23 (Estimated); Primary Completion 2025-12-23 (Estimated); Study Completion 2026-04-23 (Estimated)

PRIMARY OUTCOMES:
Change in facial skin thickness | No later than 8 weeks after the last injection
  Change from baseline in facial skin thickness following three intradermal administrations of the DensiStim product, based on ultrasound measurements.

SECONDARY OUTCOMES:
Change in facial skin thickness based on ultrasound measurements, comparison between visits | baseline, 1 month after first injection, 1 month after second injection, 1 month after third injection and 2 months post-treatment
Change in facial skin thickness based on ultrasound measurements, comparison between study arms | baseline, 1 month after first injection, 1 month after second injection, 1 month after third injection and 2 months post-treatment
Change in facial skin parameters based on multispectral skin analysis | baseline, 1 month after first injection, 1 month after second injection, 1 month after third injection and 2 months post-treatment
Change in aesthetic improvement and psychological well-being scores, assessed by participants | baseline, 1 month after first injection, 1 month after second injection, 1 month after third injection and 2 months post-treatment
Change in aesthetic improvement scores, assessed by the Investigator | baseline, 1 month after first injection, 1 month after second injection, 1 month after third injection and 2 months post-treatment
Percentage of participants satisfied with the results of the injections | 1 months and 2 months post-treatment
Post-injection sensation scores, assessed by participants using the Numeric Rating Scale Questionnaire | after first injection, after second injection, after third injection
  NRS scale 0-10, where 0 indicates no pain/stinging/burning/sensation of pressure, and 10 indicates the worst imaginable pain/stinging/burning/sensation of pressure
Incidence of adverse events by event type | From enrollment to 2 months after the last injection
Percentage of participants who discontinued treatment due to adverse events | From enrollment to 2 months after the last injection

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Sirocka, Principal Investigator
Locations (1):
- Dr Agnieszka Sirocka - Medycyna Estetyczna, Kowale, Poland